CLINICAL TRIAL: NCT04557891
Title: Feasibility of Low-Intensity Focused Ultrasound Pulsation (LIFUP) for the Treatment of Generalized Anxiety Disorder (GAD)
Brief Title: Low-Intensity Focused Ultrasound Pulsation (LIFUP) for the Treatment of Generalized Anxiety Disorder (GAD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Massachusetts General Hospital (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Margaret Distler, MD, PhD, Health Sciences Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTP-LIFUP-GAD-V1.0
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: focused ultrasound
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Low Intensity Focused Ultrasound (Experimental): Device: Low Intensity Focused Ultrasound Device
  Low Intensity Focused Ultrasound Pulsation (LIFUP) of amygdala (a key area for anxiety) will be performed during two sessions. The proposed experiment will involve behavioral (e.g. HAM-A) and paramedical (i.e., MRI/fMRI) measurements just before and after each of the two LIFUP sessions (i.e., 5 non-consecutive minutes of stimulation in each session). The device does not produce a sound when operating and as such, the active group will well blinded.
  Interventions: Device: Active LIFUP Treatment
- Sham (Sham Comparator): Sham Treatment consists of placing the device but not turning it on. The device does not produce a sound when operating and as such, the sham group will well blinded.
  Interventions: Device: Sham LIFUP Treatment

INTERVENTIONS:
Device: Active LIFUP Treatment — 8 LIFUP Treatments
  Other Names: BX Pulsar 1002
  Arms: Low Intensity Focused Ultrasound
Device: Sham LIFUP Treatment — 8 sham LIFUP treatments
  Arms: Sham

SUMMARY:
There are few treatment options available for patients once they have failed standard psychopharmacological therapy for generalized anxiety disorder. Existing brain stimulation methods such as rTMS fail to target deep brain structures associated with anxiety disorders; structures such as the amygdala. In this double-blind sham-controlled clinical trial, the investigators propose to establish baseline severity of anxiety in 48 patients, then deliver eight treatments over four sessions of focused ultrasound stimulation to the amygdala. Anxiety severity will be assessed using standard psychometric scales after each session, and at follow-ups.

DETAILED DESCRIPTION:
Anxiety disorders have tremendous disease burden in the United States. Up to 1 in 3 Americans will be diagnosed with an anxiety disorder in their lifetimes. Anxiety treatment is typically consisting of psychotherapy (e.g. cognitive behavioral therapy) and medication management (e.g. benzodiazepines, selective serotonin reuptake inhibitors, etc). With major depressive disorder, rTMS is a suitable alternative treatment for refractory depression, rTMS is not approved for treatment of anxiety, nor can rTMS stimulate deep enough to reach those brain circuits involved in anxiety (e.g. the amygdala). Focused ultrasound is a new treatment modality being developed for several different neuropsychiatric conditions. In this study, the investigators propose to randomize 48 individuals to either active or sham treatment. Each participant will be evaluated to establish a baseline diagnose of generalized anxiety disorder, and then will be reassessed after each treatment session (of which there are four). One week and one month after the last treatment session, the investigators will conduct follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18-65
3. Normal or corrected-to normal vision and hearing
4. Primary diagnosis of generalized anxiety disorder, moderate/severe per DSM-5. (HAM-A>17) 4a) The duration of the illness must exceed one year.
5. Must be medically stable as determined by investigator
6. Patient must have attempted and failed treatment with at least 2 SSRI and 1 augmentation
7. History of rTMS is permitted, but not required.

Exclusion Criteria:

1. Diagnosis of primary DSM-5 anxiety disorder other than GAD 1a) Affective disorders such as unipolar or bipolar depression are permitted as long as GAD is primary
2. Current use of any non-prescribed psychoactive medications or drugs (aside from medications for treatment of GAD)
3. Contraindication to enter the MRI environment
4. Pregnancy (or suspected/possible pregnancy or plan to become pregnant in the short-term)
5. Inability to adhere to treatment schedule
6. Initiation of new anxiolytic treatment at the time of study randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | 1 week after the fourth LIFUP treatment
  HAM-A is a rating scale for measuring the severity of anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret G Distler, MD,PhD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No